CLINICAL TRIAL: NCT00030095
Title: A Phase I Trial Of 2-Methoxyestradiol (2ME2), (NSC-659853) An Angiogenesis Inhibitor, In Patients With Solid Tumors
Brief Title: 2-Methoxyestradiol in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000069022; NCI-01-C-0256; NCI-3371; NCI-CC-01-C-0256; NCT00024609 (obsolete NCT alias)
Record Dates: First submitted 2002-01-30; First posted 2003-01-27 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2006-07

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — 2-Methoxyestradiol

INTERVENTIONS:
Drug: 2-methoxyestradiol

SUMMARY:
RATIONALE: 2-Methoxyestradiol may stop the growth of cancer by stopping blood flow to the tumor.

PURPOSE: Phase I trial to study the effectiveness of 2-methoxyestradiol in treating patients who have advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of 2-methoxyestradiol in patients with advanced solid tumors.
* Determine the side effect profile of this drug in these patients.
* Determine the pharmacokinetic profile of this drug in these patients.
* Determine the changes in positron-emission tomography scans of patients treated with this drug.
* Determine the changes in apotosis in patients treated with this drug.

OUTLINE: This is a dose-escalation study.

Patients receive oral 2-methoxyestradiol (2ME2) once on day 1 followed by 2 days of evaluation. Patients then receive oral 2ME2 every 12 hours. Treatment continues in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of 2ME2 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Patients are followed at day 30.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed solid tumor

  * Metastatic or unresectable disease for which standard curative treatments do not exist or are no longer effective
* Clinically progressive disease documented by any of the following:

  * New area of malignant disease
  * Progression of soft-tissue metastases
  * At least 1 new metastatic deposit on technetium Tc 99m bone scintigraphy
  * Increases in prostate-specific antigen
* Lesions accessible for serial biopsy
* No known brain metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2 OR
* Karnofsky 60-100%

Life expectancy:

* More than 3 months

Hematopoietic:

* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin normal
* AST/ALT no greater than 2.5 times upper limit of normal

Renal:

* Creatinine normal OR
* Creatinine clearance at least 60 mL/min

Cardiovascular:

* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia

Other:

* No other concurrent uncontrolled illness
* No ongoing or active infection
* No prior allergic reactions to compounds of similar chemical or biological composition to 2-methoxyestradiol
* No psychiatric illness or social situation that would preclude study compliance
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception for 1 month before, during, and for 1 month after study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior biologic therapy

Chemotherapy:

* At least 4 weeks since prior chemotherapy (6 weeks for mitomycin, nitrosoureas, or carboplatin)
* No concurrent chemotherapy for cancer

Endocrine therapy:

* Luteinizing-hormone releasing-hormone agonist therapy must be continued for patients with prostate cancer except those with prior orchiectomy

Radiotherapy:

* At least 4 weeks since prior radiotherapy
* No concurrent radiotherapy for cancer

Surgery:

* See Endocrine therapy

Other:

* Recovered from prior therapy
* No other concurrent therapy for cancer
* No concurrent combination antiretroviral therapy for HIV-positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-09

CONTACTS AND LOCATIONS:
Overall Officials: William Dahut, MD, Study Chair — NCI - Medical Oncology Branch
Locations (2):
- United States (2):
  - Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland
  - NCI - Center for Cancer Research, Bethesda, Maryland

REFERENCES:
- [Background] Lakhani NJ, Sarkar MA, Venitz J, Figg WD. 2-Methoxyestradiol, a promising anticancer agent. Pharmacotherapy. 2003 Feb;23(2):165-72. doi: 10.1592/phco.23.2.165.32088. PMID 12587805
- [Result] Lakhani NJ, Sparreboom A, Venitz J, et al.: Single oral dose pharmacokinetics (PK) and safety of 2-methoxyestradiol (2ME2) in patients with solid tumors. [Abstract] J Clin Oncol 23 (Suppl 16): A-2071, 152s, 2005.
- [Result] Dahut WL, Lakhani N, Kohn EC, et al.: A phase I study of 2-methoxyestradiol (2ME2) in patients with solid tumors. [Abstract] Proceedings of the American Society of Clinical Oncology 22: A-833, 2003.